CLINICAL TRIAL: NCT03897894
Title: A Randomised Control Trial of Enhanced Child Friendly Space Interventions for Girls and Boys Affected by Conflict and Displacement
Brief Title: Enhanced Child Friendly Space Interventions for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Elrha (Other); World Vision (Other)
Responsible Party: Principal Investigator, Cassie Landers, Ed.D, MPH, Assistant Professor of Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AAAS1367
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Psychosocial Stressors; Child, Only; Mental Health Wellness 1; Child Development
Keywords: resilience; child protection; child development

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Service Package (Experimental): The enhanced service package provides 40 sequential sessions selected by CFS program staff in advance and implemented over a twelve-week period. Activities are meant to build upon and reinforce one another and are organized into seven psychosocial themes: 1) Building community: "Our space together", 2) Emotional learning: "My feelings", 3) Wellbeing and coping: "Feeling good", 4) Social support: "My friends and family", 5) Relating to others: "Being a good friend", 6) Protection and boundaries: "My safety", and 7) Building on strengths: "All my supports". Each session takes approximately 1.5 - 2 hours to facilitate and will conclude with 1-1.5 hours unstructured free play time.
  Interventions: Behavioral: Child Friendly Space
- Basic Service Package (Experimental): The basic service package offers a mixture of recreational and non-formal education activities over a twelve-week period. Each session lasts around 1.5 - 3 hours. Structured activities offered include basic literacy and numeracy lessons, life skills exercises, health and hygiene sessions, and traditional song and dance. Many activities are centered around various forms of play that enable expression and age-appropriate skill development. Unstructured free play and playground time is allocated throughout the daily session.
  Interventions: Behavioral: Child Friendly Space
- Control (No Intervention): Waitlist control will receive delayed treatment of intervention after the primary assessment period.

INTERVENTIONS:
Behavioral: Child Friendly Space — Child Friendly Spaces (CFS) are one of the most widely used interventions to provide Mental Health and Psychosocial Support (MHPSS) as well as provide a protective environment for children in humanitarian settings.
  Arms: Basic Service Package; Enhanced Service Package

SUMMARY:
A 3-arm randomised controlled trial will be conducted to compare the effectiveness of a new enhanced Child Friendly Space service package with the basic Child Friendly Space service implementation, and to a waitlist control condition, within the West Nile refugee response in Uganda.

DETAILED DESCRIPTION:
A Child Friendly Space (CFS) is an acute phase humanitarian intervention designed to provide children with a safe, supportive, and stable environment early after the onset of crisis that will promote their social and emotional well-being, as well strengthen the existing systems of protection required to support children in reaching developmental milestones. Typically, CFSs house a range of structured and unstructured activities led by trained animators in a community-designated safe area.

The basic service package offers a mixture of recreational and non-formal education activities over a twelve-week period. Each session lasts around 1.5 - 3 hours. Structured activities offered include basic literacy and numeracy lessons, life skills exercises, health and hygiene sessions, and traditional song and dance. Many activities are centered around various forms of play that enable expression and age-appropriate skill development. Unstructured free play and playground time is allocated throughout the daily session.

The enhanced service package provides 40 sequential sessions selected by CFS program staff in advance and implemented over a twelve-week period. Activities are meant to build upon and reinforce one another and are organized into seven psychosocial themes: 1) Building community: "Our space together", 2) Emotional learning: "My feelings", 3) Wellbeing and coping: "Feeling good", 4) Social support: "My friends and family", 5) Relating to others: "Being a good friend", 6) Protection and boundaries: "My safety", and 7) Building on strengths: "All my supports". Each session takes approximately 1.5 - 2 hours to facilitate and will conclude with 1-1.5 hours unstructured free play time.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver has a child between the ages 6-8
* Child is between the ages of 9-14 years

Exclusion Criteria:

* No child resides in the home between the ages of 6 and 14 years

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2015 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Child and Youth Resilience Measure (CYRM-28) | up to 1 hour from the start of a session
  A 28-item caregiver (for children aged 6-8 years) or child-reported (for children aged 9-14 years) measure that explores the resources that may bolster the resilience of children. Each item of the child self-report has response options rated on a 5-point scale ranging from 1 (Not at all) to 5 (A Lot). Higher scores are indicative of increased presence of resilience processes. Each item of the caregiver-reported measure has three response options - 1 (No), 2(Sometimes), and 3 (Yes). Higher scores are indicative of increased presence of resilience processes of the child (better outcome).

SECONDARY OUTCOMES:
Child PTSD Symptom Scale (CPSS) Part 1 | up to 1 hour from the start of a session
  A two-part 27-item measure of psychological distress that maps to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Post-traumatic Stress Disorder (PTSD). Part one features 20 PTSD symptom items rated on a 5-point scale of frequency and severity from 0 (not at all) to 4 (6 or more times a week). Scores on part one range from 0 to 80, with higher scores indicating greater psychological distress (more symptoms) and lower scores indicating a better outcome. This will be administered to children aged 9 to 14 years.
Child PTSD Symptom Scale (CPSS) Part 2 | up to 1 hour from the start of a session
  A two-part 27-item measure of psychological distress that maps to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Post-traumatic Stress Disorder (PTSD). Part two features 7 dichotomous functionality items from 0 (no) to 1 (yes). Scores on part two range from 0 to 7, with higher scores indicating greater daily functional impairment. This will be administered to children aged 9 to 14 years.
Children's Hope Scale (CHS) | up to 1 hour from the start of a session
  A 6-item measure of children's perception of agency and pathways thinking towards goals. The CHS measures goal-oriented thinking using six youth-appropriate items. Each item has response options rated on a six-point Likert-type scale ranging from one (None of the Time) to six (All of the Time). Higher scores are indicative of more positive goal-oriented thinking (greater hopefulness). This will be administered to children aged 9 to 14 years. Caregivers of children aged 6 to 8 years will be asked to answer on behalf of their child.
Children's Revised Impact of Events Scale (CRIES-8) | up to 1 hour from the start of a session
  A 8-item screening measure of intrusive and avoidant cognitions related to PTSD and is frequently used in evaluating stress reactions after traumatic experiences. Response options are rated on a 4-point scale from 1 (Not at all) to 4 (Often). Scores range from 8 to 32, with higher scores indicating PTSD symptoms consistent with intrusion and avoidance of the child and lower scores indicating lesser PTSD symptoms (better outcome). This will be administered to caregivers of children aged 6 to 8 years.
Short Mood and Feelings Questionnaire (S-MFQ) | up to 1 hour from the start of a session
  A 13-item screening measure for depression. Each item is rated on a 3-point Likert scale with response options of 0 (Not True), 1(Sometimes True), and 2 (True). Scores range from 0 to 26, with lower scores indicating the child is likely not suffering from depression (better outcome). This will be administered to caregivers of children aged 6 to 8 years.
Emergency Developmental Assets Profile (EMDAP) | up to 1 hour from the start of a session
  A 13-item measure of developmental assets essential for children to thrive into adulthood. Each item is answered on a four-point scale from 0 (Not at All/Rarely) to 3 (Extremely/Almost Always). Scores range from 0 to 30, with higher scores indicating the child has more developmental assets (better outcome). This will be administered to children aged 9 to 14 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cassie Landers, PhD, Principal Investigator — Columbia University
Locations (1):
- World Vision West Nile Response Office, Arua, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metzler J, Saw T, Nono D, Kadondi A, Zhang Y, Leu CS, Gabriel A, Savage K, Landers C. Improving adolescent mental health and protection in humanitarian settings: longitudinal findings from a multi-arm randomized controlled trial of child-friendly spaces among South Sudanese refugees in Uganda. J Child Psychol Psychiatry. 2023 Jun;64(6):907-917. doi: 10.1111/jcpp.13746. Epub 2023 Jan 2. PMID 36593181
- See also: Project description on Donor Website — https://www.elrha.org/project/randomised-control-trial-of-enhanced-child-friendly-space-interventions-for-girls-and-boys-affected-by-conflict-and-displacement/